CLINICAL TRIAL: NCT04782986
Title: Pan-intestinal Capsule Endoscopy Versus Conventional Colonoscopy in Iron Deficiency Anemia or Overt GI Bleeding: a Prospective Cohort Study
Brief Title: Pan-intestinal Capsule Endoscopy Versus Colonoscopy in Iron Deficiency Anemia or Overt GI Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unidade Local de Saúde do Alto Ave, EPE (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Bruno Rosa, MD, Unidade Local de Saúde do Alto Ave, EPE
Allocation: Non-Randomized | Model: Factorial | Masking: Double | Purpose: Diagnostic
Other Study IDs: ERP-2020-12296
Record Dates: First submitted 2021-02-20; First posted 2021-03-04 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Iron Deficiency Anemia; GastroIntestinal Bleeding
Keywords: iron deficiency anemia; gastrointestinal bleeding; pan-intestinal capsule endoscopy
MeSH Terms: conditions — Anemia, Iron-Deficiency; Gastrointestinal Hemorrhage | interventions — Endoscopy

STUDY DESIGN:
Intervention Model Description: Prospective, single-blinded, single center cohort study. All patients will undergo pan-intestinal capsule endoscopy followed by conventional colonoscopy with deep sedation in the same day, with no need for further bowel preparation.
Who Masked: Care Provider, Investigator
Masking Description: The capsule endoscopy reader will be independent from the physicians performing the conventional colonoscopies, and all investigators will be blinded to each other's findings and reports. Capsule endoscopy and colonoscopy findings will be compared and in case of disagreement it will be discussed until a consensus is reached, if necessary, with the intervention of an independent third reader, experienced in both techniques and not involved in the primary reading of any of the examinations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pan-intestinal capsule endoscopy (Experimental): PillCam Crohn's capsule protocol
  Interventions: Diagnostic Test: Pan-intestinal capsule endoscopy
- Conventional colonoscopy (Active Comparator): Same-day colonoscopy under propofol sedation
  Interventions: Diagnostic Test: Pan-intestinal capsule endoscopy

INTERVENTIONS:
Diagnostic Test: Pan-intestinal capsule endoscopy — Patients with iron deficiency anemia or overt GI bleeding with non-diagnostic upper GI endoscopy will be submitted to same-day pan-intestinal capsule endoscopy using PillCam Crohn's Capsule (Medtronic) followed by conventional colonoscopy under propofol sedation
  Other Names: Conventional colonoscopy

SUMMARY:
The authors hypothesize that in patients with iron deficiency anemia or gastrointestinal bleeding, pan-intestinal capsule endoscopy is a safe and well tolerated procedure that may improve diagnostic yield comparatively to the current standard invasive colonoscopy.

DETAILED DESCRIPTION:
Patients presenting with iron deficiency anemia (IDA) or overt GI bleeding are often submitted to conventional upper GI endoscopy and colonoscopy, followed by small bowel capsule endoscopy if diagnosis remains elusive. Recently, however, the possibility of performing pan-intestinal endoscopy using a video capsule that evaluates both the small bowel and the colon in a single non-invasive examination, opens new perspectives for the management of those conditions, particularly when the initial upper GI endoscopy has been non-diagnostic. The authors hypothesize that performing early pan-intestinal capsule endoscopy strategy may allow, in a safe and well tolerated manner, to identify which patients would benefit of further interventions, such as colonoscopy or invasive enteroscopy, guided by findings pre-identified at capsule examination. The study aims to evaluate whether pan-intestinal capsule endoscopy is superior to the current standard strategy of conventional colonoscopy after non-diagnostic upper endoscopy in patients with IDA or overt GI bleeding, regarding diagnostic yield, safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Patients from external consultation, hospital ward or urgency department, with suspected GI bleeding presenting in the occult form as IDA (Hb <12.0 g/dL in female gender or <13.0 g/dL in male gender) and/or overt GI bleeding presenting as melaena and/or haematochezia, and with prior non-diagnostic upper GI endoscopy (esophagogastroduodenoscopy, EGD)

Exclusion Criteria:

1. Lack of informed consent
2. Suspected lesions at index EGD that could justify the anemia or digestive bleeding
3. Known history of gastroparesis or bowel dysmotility
4. Known or suspected intestinal stricture
5. Female patients with potential gynaecological source of bleeding causative of the clinical condition
6. Patients with severe malnutrition
7. Patients unable to walk at least for short periods and/or with neurological and/or psychiatric condition potentially favouring protocol deviations
8. Allergy or contra-indications to any of the drugs or products used in the study
9. Pregnancy or breastfeeding

Ages: 8 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with at least one potentially bleeding lesion detected in small bowel and/or colon | 2 weeks
  Potentially bleeding lesions include tumors, angiectasias, erosions, ulcers, diverticula or active bleeding

SECONDARY OUTCOMES:
Safety: number of participants with any procedure-related adverse events | 2 weeks
  Adverse events include capsule retention, bowel preparation-related (nausea, vomiting, dizziness, seizures, abdominal pain or bloating), bleeding, perforation or cardiopulmonary complications
Patient's preference: number of participants preferring capsule endoscopy or colonoscopy | 2 weeks
  Questionnaire regarding preference based on overall experience and perception of the strengths and limitations of each procedure

OTHER OUTCOMES:
Quality of bowel preparation at capsule endoscopy (small bowel) | 2 weeks
  Use of validated Brotz scale (4-grade qualitative assessment as excellent, good, fair or poor bowel preparation)
Quality of bowel preparation at capsule endoscopy (colon) | 2 weeks
  Use of validated scale CC-CLEAR (Colon Capsule CLEansing Assessment and Report) - quantitative scale: adequate bowel preparation if overall score >= 6 points, and >= 2 points in each bowel segment (right, transverse, and left colon). Overall 0-5 points inadequate; 6-7 points good; 8-9 points excellent bowel preparation
Quality of bowel preparation at colonoscopy | 2 weeks
  Use of validated Boston Bowel Preparation Scale: quantitative scale 0-9 points - adequate bowel preparation if overall score >= 6 points, and >= 2 points in each bowel segment (right, transverse, and left colon)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Rosa, MD, Principal Investigator — Gastroenterology Department, Hospital da Senhora da Oliveira - Guimarães, Portugal
Locations (1):
- Gastroenterology Department, Hospital da Senhora da Oliveira, Guimarães, Portugal

IPD SHARING:
Plan to Share IPD: No